CLINICAL TRIAL: NCT01584466
Title: Long Acting Paliperidone in Dually Diagnosed People With Schizophrenia: An Open-label Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Heidi Wehring, PharmD, BCPP, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00052194
Record Dates: First submitted 2012-03-20; First posted 2012-04-25 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Substance Abuse
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone (Experimental)
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — The starting regimen will be a 'loading dose' strategy whereby the first injection will be 234 mg given on treatment week 0,day 1 and 156 mg (2nd injection) will be given 1 week later (days 5-9). Both are recommended to be administered in the deltoid muscle (PI 2011). Following the second dose, monthly maintenance doses will be administered in either the deltoid or gluteal muscle (PI 2011). The monthly (± 7 days) maintenance dose will be 117 mg.
  Discontinuation of oral antipsychotics is recommended after the subjects receive paliperidone palmitate injection on Week 0/day 1. Continued oral antipsychotics may be used only if necessary.

SUMMARY:
Comorbid substance abuse leads to many deleterious effects such as medical comorbidities and nonadherence, which is one of the most problematic issues. People with schizophrenia and substance use disorders (SUDs) are at an increased risk nonadherence compared to those who do not use alcohol and illicit drugs. The investigators propose that this new marketed injectable antipsychotic with many benefits over other available long acting injectable agents would be beneficial in the dually diagnosed population and may represent a specific schizophrenia subpopulation where long acting agents may be considered an important therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 18 and 64
* Either gender
* Any race
* Meet DSM-IV-TR criteria for Schizophrenia or Schizoaffective Disorder.
* Alcohol and/or cannabis use defined as a DSM-IV diagnosis abuse, dependence or regular use defined as 3 times per week during the past year
* Agree to take or use birth control during the study.

Exclusion Criteria:

* Previous lack of response or serious adverse event to risperidone or paliperidone.
* Currently on a long acting injectable antipsychotic.
* A score of less than 10 on the Evaluation to Sign Consent (ESC).
* Medical illnesses, which may compromise safe study participation.
* Pregnant and lactating females.
* QTc interval > 450 milliseconds males or > 470 milliseconds in females
* Currently on acamprosate, naltrexone and disulfiram.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Long acting paliperidone palmitate will improve psychotic, negative and depressive symptoms from baseline to endpoint | 7 months
  Long acting paliperidone palmitate will improve psychotic, negative and depressive symptoms from baseline to endpoint during six months of treatment. Improvement in psychotic symptoms will be measured by decrease in the Brief Psychiatric Rating Scale (BPRS) psychosis score. Improvement in negative symptoms will be measured by decrease in the Scale for the Assessment of Negative Symptoms (SANS) total score. Improvement in depressive symptoms will be measured by decrease in Calgary Depression Scale (CDS) total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States